CLINICAL TRIAL: NCT02595736
Title: A Single Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of LY3200327 in Healthy Subjects
Brief Title: A Study of LY3200327 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 15577; I8C-MC-GSFA (Other: Eli Lilly and Company)
Record Dates: First submitted 2015-11-02; First posted 2015-11-03 (Estimated); Last update posted 2016-09-12 (Estimated); Status verified 2016-09

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo (SC) (Placebo Comparator): Single subcutaneous (SC) dose of placebo
  Interventions: Drug: Placebo (SC)
- LY3200327 (SC) (Experimental): Single escalating subcutaneous (SC) dose of LY3200327
  Interventions: Drug: LY3200327 (SC)
- LY3200327 (IV) (Experimental): Single intravenous (IV) dose of LY3200327
  Interventions: Drug: LY3200327 (IV)
- Placebo (IV) (Placebo Comparator): Single intravenous (IV) dose of placebo
  Interventions: Drug: Placebo (IV)

INTERVENTIONS:
Drug: Placebo (SC) — Administered SC
  Arms: Placebo (SC)
Drug: LY3200327 (SC) — Administered SC
  Arms: LY3200327 (SC)
Drug: LY3200327 (IV) — Administered IV
  Arms: LY3200327 (IV)
Drug: Placebo (IV) — Administered IV
  Arms: Placebo (IV)

SUMMARY:
The purpose of this study is to look at the safety and tolerability of single doses of LY3200327 when given to healthy male and female participants either by injection under the skin or by drip into a vein. The study will help determine how the drug behaves inside the body and how long it takes to disappear from the body. The study will also look for anti-drug antibodies and how these may affect how LY3200327 acts in your body.

The study is expected to last approximately 12 weeks (with screening evaluations up to 4 weeks prior).

ELIGIBILITY:
Inclusion Criteria:

* At the time of initial screening, in general good health
* First-generation healthy Japanese (age 20 to 65 years) will be included

Exclusion Criteria:

* Pregnancy or breastfeeding during the study
* Chronic infection
* Treatment with prohibited medications

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2015-11; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Number of Participants with One or More Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to Study Drug Administration | Baseline to study completion (approximately 12 weeks)

SECONDARY OUTCOMES:
Pharmacokinetics (PK): Maximum Concentration (Cmax) of LY3200327 | Pre-dose up to 84 days post dose
Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve (AUC) of LY3200327 | Pre-dose up to 84 days post dose

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Parexel International/ California Clinical Trials, Glendale, California, United States